CLINICAL TRIAL: NCT05506839
Title: A Scalable Model for Promoting Functioning and Well-Being Among Veterans With a History of Mental Health Challenges Via Meaningful Social Interactions: Project V-SPEAK!
Acronym: V-SPEAK!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, Professor of Health Behavior and Health Education, and of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00216275
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Depression, Anxiety; PTSD
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Participants will be paired with an English language learner and engage in 8 weeks, 1 hour videoconferencing sessions.
  Interventions: Other: Intervention (videoconferencing)

INTERVENTIONS:
Other: Intervention (videoconferencing) — 1 hour videoconferencing sessions over 8 weeks with an English language learner partner.

SUMMARY:
The goal of this study is to refine and test a strategy for engaging veterans with symptoms of depression and/or anxiety as volunteers to help English language learners (ELLs) improve their speaking skills via structured conversations using videoconferencing.

DETAILED DESCRIPTION:
The program to be refined and pilot tested is called V-SPEAK! - Veteran Service Promoting English Acquisition and Knowledge. Through V-SPEAK!, veterans with a history of mental health concerns will volunteer as coaches, helping English Language Learners (ELL) improve their verbal English skills via structured conversations using webcams. In August 2018, there was a focus group with veterans, including both genders, African Americans, and veterans with challenges such as generalized anxiety disorder, post-traumatic stress disorder, and depression. The group universally felt that V-SPEAK! fit well with veterans' sense of service and could be beneficial for those struggling with a loss of purpose, loneliness, and decreased self-worth. Veterans with mental disorders mentioned that the structured, bounded interactions via webcam would be an ideal way to increase social engagement without triggering anxiety or feeling overwhelmed.

The proposed study is designed to provide initial pilot data on the potential feasibility and impact of V-SPEAK! for veterans who have had mood disorders. Based on this study, there will be further refinement of the program and, if the results are positive, the investigator will seek grant funding for a more rigorous evaluation of the program's impact on outcomes. Despite the extremely encouraging experience to date recruiting participants for other similar studies (e.g., older adult volunteers with mild cognitive impairment), an important goal will be to determine whether the study can recruit and retain veterans with depression or anxiety, as well as the ELL conversation partners. Also the current V-SPEAK! orientation and session-support materials will be tailored to address the unique needs of veterans, and preliminary data on satisfaction with the V-SPEAK! experience and its impact on participants' mental health and functioning will be gathered. The study will provide vital data for the submission of a competitive application for a larger randomized trial evaluating the intervention's impact on veterans' mental health (e.g., depression, loneliness, and sense of purpose).

ELIGIBILITY:
Veteran coach participant --

Inclusion Criteria:

* 18 years of age or older
* fluent English speakers
* be able to participate in a videoconference via a smartphone, tablet, laptop, or desktop computer in their home using a widely-accessible, no cost videoconferencing platform.

Exclusion Criteria:

* schizophrenia
* dementia
* traumatic brain injury
* significant sensory impairment
* current alcohol or drug abuse/dependence that would affect their ability to participate in the study

English Language Learner participant --

Inclusion Criteria:

* 18+ years of age
* be able to participate in a videoconference via a smartphone, tablet, laptop, or desktop computer in their home or referring organization using a widely-accessible, no cost videoconferencing platform
* basic ability to understand and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  The Psychological Wellbeing Scale (PWB) is a validated measure shown to be sensitive to intervention effects. This is a 6 point scale where the minimum is 1 (strongly disagree) and maximum is 6 (strongly agree). Higher scores reflect higher wellbeing.
France and Finney "Mattering" | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  This is a 5 point scale where the minimum is 1 (strongly disagree) and maximum is 5 (strongly agree). Higher scores reflect higher mattering, and mattering is positively related to measures of well-being.
Brief Inventory of Thriving | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  This is a 5 point scale (1=strongly disagree to 5=strongly agree). Higher scores reflect a greater sense of well-being.
3-item UCLA (University of California, Los Angeles) Revised Loneliness Scale | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  This is a 3 point scale from 1=hardly ever to 3=often (minimum is 1 maximum is 3). The scores for each individually answered questions can be added together to give you a possible range of scores from 3-9. Score of 3-5 is "not lonely" and score of 6-9 is "lonely".
(Patient Health Questionnaire) PHQ-8 | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  This is a 3 point scale (0= not at all, 3= nearly every day). Higher scores reflects greater depression.
(Generalized Anxiety Disorder) GAD-7 | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  This is a 3 point scale (0= not at all, 3= nearly every day). Higher scores reflects greater anxiety.
(Posttraumatic Stress Disorder Checklist) PCL-5 | Baseline and Follow-up (administered after the 8 weekly conversation sessions)
  PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. 5-point Likert (0 = "Not at all" to 4 = "Extremely"). Research on the PCL-5 suggested scores of 31 to 33 were optimally efficient for diagnosing PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, North Campus Research Complex, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT05506839/ICF_000.pdf